CLINICAL TRIAL: NCT05961449
Title: Disentangling Peripheral and Central Mechanisms of Exercise-induced Hypoalgesia in Healthy Adults Males.
Brief Title: Mechanisms of Exercise-induced Hypoalgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: EIH
Record Dates: First submitted 2023-07-06; First posted 2023-07-27 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Healthy; Men; Adults
Keywords: healthy; males; adults
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Intervention Model Description: A within-subject, cross-over design, will be used: participants will complete two conditions (exercise vs. control) in counter-balanced randomized order.
Who Masked: Participant
Masking Description: Participants will be blinded to the study hypotheses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental condition (Experimental): Participants will complete an experimental exercise that will consist in 25 minutes of cycling between 60-80 Revolution Per Minute (RPM) on a cycle ergometer (CST BX40; Cardiostrong; Germany) at ≥ 70% of the Heart Rate Reserve (HRR).
  Interventions: Behavioral: Cycling exercise
- Control condition (Sham Comparator): The control condition will include an exercise design similar to the experimental condition except that the resistance will be kept at 25 W and the RPM below 50. The intensity of the exercise will be kept at minimal levels by ensuring that the heart rate does not increase >25% from baseline
  Interventions: Behavioral: Cycling control

INTERVENTIONS:
Behavioral: Cycling exercise — Participants will complete an experimental exercise that will consist in 25 minutes of cycling between 60-80 Revolution Per Minute (RPM) on a cycle ergometer (CST BX40; Cardiostrong; Germany) at ≥ 70% of the Heart Rate Reserve (HRR).
  Arms: Experimental condition
Behavioral: Cycling control — The control condition will include an exercise design similar to the experimental condition except that the resistance will be kept at 25 W and the RPM below 50. The intensity of the exercise will be kept at minimal levels by ensuring that the heart rate does not increase >25% from baseline.
  Arms: Control condition

SUMMARY:
This project aims to clarify the mechanisms underpinning the acute analgesic effect of exercise in healthy humans-a phenomenon called "Exercise-induced hypoalgesia" (EIH). This study will characterize, using a within-subject cross-over design, the effects of a single session of aerobic exercise vs. a control condition on the sensitivity to stimuli preferentially activating mechano vs. heat-sensitive nociceptors of the skin vs. muscle, within vs. outside exercising body parts. The investigators hypothesize (1) that EIH will be greater in the exercise session compared to the control session, (2) that EIH will be greater at the local site compared to the remote site if local changes in nociceptive sensitivity contribute to EIH, and (3) that exercise will preferentially affect blunt pressure-induced pain if EIH involves specific changes in sensitivity of muscle nociceptors.

ELIGIBILITY:
Inclusion Criteria:

* Males aged between 18 and 30 years
* Lack of risks for physical exercise assessed using the Physical Activity Readiness Questionnaire (PAR-Q)
* Ability to provide written informed consent
* Fluency in French
* BMI between 17 and 30

Exclusion Criteria:

* Regular tobacco use
* Not willing or able to abstain from alcohol, recreational drugs, coffee, or tea from 24 hours prior to each experimental session.
* Not willing or able to restrain from physical activity > 24h prior to each experimental session, and to be in a fasted state on the day of each experimental session.
* Any neurological, cardio-vascular, respiratory, inflammatory, endocrine, psychiatric, oncological, rheumatological conditions. Such condition could put the participants at risk during maximal exercise testing and/or interfere with pain assessment.
* Presence of any medical devices (e.g., cardiac pacemaker) implants or prothesis unless it is beyond discussion that these will not put the subject's safety during the study at risk and will not interfere with the results of the study.
* Any chronic pain condition or recent history thereof (i.e. within the preceeding 2 years).
* Wounds or skin alteration on testing sites.
* Impaired hearing. This would affect ability to detect the control auditory stimuli.
* Surgery < 12 months
* Any drug intake in the past 2 weeks including antibiotics, herbal medicines and other remedies except the following drugs that will be allowed up to 48 hours prior to the experiments: oral paracetamol or ibuprofen for a self-limiting condition (e.g. toothache, bruise). Oral antihistaminics and nasal aerosol and topical treatments for seasonal allergy up to 1 week before the experimental session.
* Any physical activity contraindication

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Change in pressure pain threshold | Throughout the entire study, approximately during 6 months
  The investigators will use blunt pressure to preferentially activate the mechano-sensitive deep-tissue nociceptors. The stimuli will be delivered with a manual digital algometer with a contact surface area of 1cm2 (FPIX; Wagner Instruments, Greenwich, USA) connected to a laptop computer through a USB-serial port. A bespoke Matlab (The Mathworks, USA, mathworks.com) script will provide visual feedback of the force application rate to the examinator. The participants will be asked to report the first onset of pain by pressing on a keyboard key. The procedure is safe, and there are no side effects to the stimulation. This outcome will measured before and after each of the condition of the study (experimental exercise vs. control exercise)-relative and absolute change will then be computed.
Change in cold detection threshold and heat pain threshold | Throughout the entire study, approximately during 6 months
  The investigators will apply thermal stimuli to the skin to activate selectively heat-sensitive Aδ- and C-cutaneous fibre afferents. The thermal stimuli will be produced by a contact thermode based on Peltier elements (TCS-2; QST.lab, Strasbourg). The cold detection threshold (CDT) will be estimated by asking participants to press a button as soon as a decrease in skin temperature is noticed. The heat pain threshold (HPT) will be estimated by asking participants to press a button as soon as the increase in skin temperature becomes painful. This device is safe and routinely used for diagnostic purposes. The thermal stimulators will be used, in accordance with safety guidelines. If requested by the participant, the stimulation procedure can be stopped at any time, with no after effect. This outcome will measured before and after each of the condition of the study (experimental exercise vs. control exercise)-relative and absolute change will then be computed.
Change in rating of mechanical activation of cutaneous nociceptive afferents | Throughout the entire study, approximately during 6 months
  The investigators will use calibrated mechanical pinprick stimulators with a small surface probe to selectively activate the skin mechanosensitive nociceptors (The PinPrick; MRC Systems GmbH, Heidelberg, Germany). Upon each stimulation, the participants will be asked to provide a rating of pain on a 100mm Visual Analogue Scale (VAS) anchored from "No sensation" to "Worst pain imaginable" with a mark in the middle denoting the transition from unpainful to painful sensations. To avoid sensitization/habituation of the skin, the location of the stimulus will be slightly changed for each stimulation. The sensation perceived by pinprick stimulation are most often described as pricking and sometimes like a touch sensation. The procedure is safe, and there are no side effects to the stimulation. This outcome will measured before and after each of the condition of the study (experimental exercise vs. control exercise)-relative and absolute change will then be computed.
Change in auditory detection threshold | Throughout the entire study, approximately during 6 months
  The auditory stimulation will consist in a progressively increasing tone delivered at a comfortable hearing level using a pair of commercially available headphones. The participants will report the perception of the sound by pressing on a keyboard key. This outcome will measured before and after each of the condition of the study (experimental exercise vs. control exercise)-relative and absolute change will then be computed.

CONTACTS AND LOCATIONS:
Overall Officials: André Mouraux, Full professor, MD, Principal Investigator — Institute of Neuroscience, UCLouvain
Locations (1):
- Institute of Neuroscience, UCLouvain, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No